CLINICAL TRIAL: NCT01531296
Title: Correlation Between MRI and Clinical Measurements of Lower Extremity Rotational Profile: Reliability of MRI to Assess Rotation for Femoral Version and Tibial Torsion
Brief Title: To Assess Rotation for Femoral Version and Tibial Torsion
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stephen Aoki, M.D., University of Utah
Other Study IDs: 51477
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Rotational Malalignment of the Lower Extremity
Keywords: MRI; Lower Extremity Rotational; Femoral Version; Tibial Torsion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Determining the investigators ability to accurately assess rotational malalignment clinically compared to imaging.

DETAILED DESCRIPTION:
The objectives of this study are 1) to assess the inter/intra-observer reliability of rotational measurements on axial MRI images and 2) determine the correlation between clinical and MRI measures of femoral version and tibial torsion.

The investigators will use previously obtained MRI images to retrospectively calculate the inter-observer and intra-observer reliability of our measurements. Participating physicians will undergo training to standardize measurement technique. Five orthopaedic surgeons and one radiologist will perform the measurement to calculate inter-observer reliability. To asses intra-observer reliability, repeat measurements will be performed by the same physicians at a later date (at least 2 weeks). The physicians will be blinded to previous results when performing the second set of measurements. A standardized rotational profile will be performed on all patients presenting to the investigators with patellofemoral complaints or rotational abnormalities warranting intervention. Internal and external hip rotation will be measured in the prone and supine positions. Tibial torsion will be assessed with the thigh-foot axis in the prone and sitting positions. Investigators will participate in a formal training session prior to data collection to normalize measurements. Each study participant will undergo MRI imaging of the femur and tibia.

ELIGIBILITY:
Inclusion Criteria: Retrospective:

* Prior study MRI images available in the University PACS system
* Prior study MRI images obtained at PCMC and uploaded into the OsiriX software (OsiriX is a software program compatible with multiple imaging formats that has easily adaptable measurement tools)
* We will search our imaging database from 2009 to current. Included will be all gun site MRI studies obtained at PCMC or the UOC for evaluation of rotational profile. We will exclude any study in which images are not sufficient to obtain all of the required measurements needed for our study. A preliminary review of the imaging database has identified 42 potential studies. Our power analysis calls for 15 patients to be included to obtain a 95% confidence interval.

Inclusion Criteria: Prospective:

* All patients of the investigating physicians, male and female, between the ages of 8 and 30 presenting with complaints of patellofemoral pain/instability or rotational abnormality
* All patients with neuromuscular disease, including cerebral palsy

Exclusion Criteria: Retrospective:

* Any patients with imaging studies insufficient to provide all of the required measurements and any patient previously surgically treated for rotational malalignment

Exclusion Criteria: Prospective:

* Any patient that has undergone previous surgical treatments for rotational malalignment.
* Any patients with implantable devices not compatible with MRI

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study is aiming to recruit all patients with complaints of patellofemoral pain/instability associated with rotational malalignment. The two types of rotational malalignment, fibial version and tibial torsion are most common among the pediatric population.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To assess the inter/intra-observer reliability of rotational measurements on axial MRI images | 4 years

SECONDARY OUTCOMES:
To determine the correlation between clinical and MRI measures of femoral version and tibial torsion. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aoki, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States